CLINICAL TRIAL: NCT01282944
Title: Encouraging Walking in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 812090; RC2AG036592 (NIH)
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-02

CONDITIONS: Physical Activity
Keywords: physical activity in adults 65 or older
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Combined Financial Incentive & Peer Network Arm (Experimental): Daily use of pedometer for 6 months. Walking goal set based on level of walking during 2 week run-in period. Subjects connected with 4 other participants in the same study arm to form a peer network of 5 individuals. Each peer network participant given access to a secure online message board that will allow the 5 participants in each peer network to communicate online. Participants also receive weekly feedback regarding which participants in the peer group achieved their walking goals during the previous week.
  Each week, if pedometer is used and walking goal is met for 5 out of 7 days, participant will be entered in lottery with an approximate 3 in 10 chance of winning $50 and an approximate 3 in 100 chance of winning $200.
  Financial incentive and peer network terminated after 4 months. Daily use of pedometer continues for an additional 2 months.
  Interventions: Behavioral: Financial Incentive; Behavioral: Peer Network
- Active Control (No Intervention): Daily use of pedometer for 6 months. Walking goal set based on level of walking during 2 week run-in period. Weekly feedback provided on meeting walking goal - defined as achieving goal number of steps for 5 of 7 days per week.
  Subjects in the Control Group will only receive pedometers and weekly feedback on their performance through the same mechanisms and with the same frequency as participants in the other three study arms. There will be no financial incentives or peer networks in this group.
- Financial Incentive Arm (Experimental): Daily use of pedometer for 6 months. Walking goal set based on level of walking during 2 week run-in period. Weekly feedback provided on meeting walking goal - defined as achieving goal number of steps for 5 of 7 days per week. Each week, if pedometer is used and walking goal is met for 5 out of 7 days, participant will be entered in lottery with an approximate 3 in 10 chance of winning $50 and an approximate 3 in 100 chance of winning $200. Financial incentive is terminated after 4 months. Daily use of pedometer continues for an additional 2 months.
  Interventions: Behavioral: Financial Incentive
- Peer Network Arm (Experimental): Daily use of pedometer for 6 months. Walking goal set based on level of walking during 2 week run-in period.
  Weekly feedback provided on meeting walking goal - defined as achieving goal number of steps for 5 of 7 days per week.
  Subjects will be connected with 4 other participants in the same study arm to form a peer network of 5 individuals. Each peer network participant will be given access to a secure online message board that will allow the 5 participants in each peer network to communicate online. All participants in a peer network will receive a list of ways in which his or her new network could support each individual's walking goals. Participants will also receive weekly feedback regarding which participants in the peer group were successful in achieving their walking goals during the previous week.
  Peer network is terminated after 4 months. Daily use of pedometer continues for an additional 2 months.
  Interventions: Behavioral: Peer Network

INTERVENTIONS:
Behavioral: Financial Incentive — Lottery with an approximate 3 in 10 odds of earning $50 and an approximate 3 in 100 odds of earning $200.
  Arms: Combined Financial Incentive & Peer Network Arm; Financial Incentive Arm
Behavioral: Peer Network — Subjects will be connected with 4 other participants in the same study arm to form a peer network of 5 individuals.
  Arms: Combined Financial Incentive & Peer Network Arm; Peer Network Arm

SUMMARY:
The goal of this pilot randomized controlled trial is to evaluate whether financial incentives and peer networks delivered through a novel computer platform utilizing a digital pedometer-internet interface can effectively encourage sustained increases in walking among older adults.

DETAILED DESCRIPTION:
This pilot study is a randomized controlled trial of incentive schemes delivered through a novel internet-based platform to promote walking in older adults. The four arms consist of the following: financial incentives, peer network, combined arm (financial incentive & peer network), and control.

Participation in the study will last approximately 26 weeks, including the 2-week run-in period, 4-month intervention period, and 2-month follow-up period.

The primary goals of the study are:

1. To test the effects of financial incentives on older adults uptake and retention of increased levels of walking.

   Hypothesis1a: Participants receiving financial incentives will increase their number of steps per day more than participants not receiving financial incentives.
2. To test the effects of connection to a new peer network on older adults uptake and retention of increased levels of walking.

   Hypothesis 2a: Participants connected to a new peer network of other participants will increase their number of steps per day more than participants not connected to a new network.

   Hypothesis 2b: Participants connected to a new peer network of other participants will retain increases in their number of steps per day more than participants not connected to a new network.
3. To test the combined effects of financial incentives and peer networks on older adults' uptake and retention of increased levels of walking.

   Hypothesis 3a: Participants who receive financial incentives and are connected to a peer network will increase their number of steps per day more than participants who are only connected to a peer network.

   Hypothesis 3b: Participants who receive financial incentives and are connected to a peer network will more effectively maintain increases in number of steps per day as compared with participants who only receive financial incentives.
4. To develop internet, text and email messaging, and pedometer-internet interface technologies to build peer networks and provide regular feedback to subjects.

Hypothesis 4: The study platform will provide an effective mechanism for subject recruitment, data collection, communication and regular feedback.

ELIGIBILITY:
Inclusion Criteria:

* Adult 65 years of age or older
* Communicates primarily in English
* Personal computer with high-speed internet connection and functional Universal Serial Bus (USB) port
* Able to walk 1/4 mile (i.e., 2 to 3 blocks) without stopping
* Currently engaging in less than 150 minutes moderate intensity exercise & less than 75 minutes vigorous intensity exercise each week
* No pedometer use in last 30 days
* Planning to stay in area for study duration

Exclusion Criteria:

* Myocardial infarction, stroke, transient ischemic attack, major cardiovascular surgery, deep venous thrombosis, or pulmonary embolus in the last 6 months
* New York Heart Association Class III or IV heart failure; severe aortic stenosis; history of cardiac arrest, use of cardiac defibrillator; or severe angina
* Hip fracture, total hip replacement, total knee replacement or spinal surgery in the last 6 months
* Uncontrolled hypertension
* Lung disease requiring supplemental oxygen
* Diabetes mellitus requiring insulin therapy
* Severe osteoarthritis or rheumatoid arthritis
* End stage renal disease requiring hemodialysis
* Movement disorder (e.g., Parkinson's disease)
* Dementia (e.g., Alzheimers Disease, Lewy-Body Dementia, Multi-Infarct Dementia, Picks Disease, Binswangers Disease, Frontotemporal Dementias, Parkinsons Disease Dementia, Huntingtons Disease, Dementia in HIV/AIDS, Wernicke-Korsakoff syndrome, Creutzfeldt-Jakob disease)
* Major psychiatric disorder (e.g., schizophrenia or bipolar disorder)
* Current consumption of ≥ 14 alcoholic drinks per week

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
mean proportion of days that step per day goals were attained | 16 weeks

SECONDARY OUTCOMES:
mean number of steps per day | 16 weeks
mean proportion of days that step per day goals were attained during follow-up | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jason Karlawish, MD, Principal Investigator — University of Pennsylvania; Jeffrey T Kullgren, MD, MPH, Study Director — kullgren@mail.med.edu
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States